CLINICAL TRIAL: NCT01012310
Title: A Double Blind, 3rd Party Open, Placebo Controlled, Dose Escalating, Parallel Group Study To Investigate The Safety, Toleration And Pharmacokinetics Of Multiple Oral Doses Of PF-04531083 In Healthy Subjects
Brief Title: Group Study To Investigate The Safety, Toleration And Pharmacokinetics Of Multiple Oral Doses Of PF-04531083 In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1351002
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2010-04

CONDITIONS: Healthy Volunteers
Keywords: pharmacokinetics safety tolerability multiple dosing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental)
  Interventions: Drug: PF-04531083 or Placebo
- Cohort 2 (Experimental)
  Interventions: Drug: PF-04531083 or Placebo
- Cohort 3 (Experimental)
  Interventions: Drug: PF-04531083 or Placebo
- Cohort 4 (Experimental)
  Interventions: Drug: PF-04531083 or Placebo

INTERVENTIONS:
Drug: PF-04531083 or Placebo — Subjects will receive multiple oral doses of less than or equal to 100mg PF-04531083 or placebo for 14 days.
  Arms: Cohort 1
Drug: PF-04531083 or Placebo — Subjects will receive multiple oral doses of less than or equal to 300mg PF-04531083 or placebo for 14 days.
  Arms: Cohort 2
Drug: PF-04531083 or Placebo — Subjects will receive multiple oral doses of less than or equal to 500mg PF-04531083 or placebo for 14 days.
  Arms: Cohort 3
Drug: PF-04531083 or Placebo — A fourth cohort may be used to investigate alternative dosing regimens, formulations or food effects.
  Arms: Cohort 4

SUMMARY:
The purpose of this study is to determine the safety and toleration of single and multiple doses of PF-04531083. (To investigate the plasma and urinary pharmacokinetics of PF-04531083 and its metabolites, following single and multiple dose administration in healthy male and/or female subjects; and to determine whether PF-04531083 raises levels of enzymes involved in metabolism of other drugs following multiple dosing).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects btween the ages of 18-55 years
* Body Mass Index (BMI) of 15.5 to 30.5 and a total body weight greater than 50kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically signifcant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 21 drinks/week within 6 months of screening
* Use of tobacco or nicotine containing products in excess of the equivalent of 5 cigarettes per day.
* Pregnant or nursing females; females of childbearing potentioal who are unwilling or unable to use an acceptable method on contraception.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of PF-04531083 Cmax, Tmax, AUCtau, AUCinf, T1/2, accumulation index | days 1-15
Safety of subjects following multiple dosing of PF-04531083 (adverse events, vital signs measurements, telemetry, 12-lead ECGs, physical examination findings, blood and urine safety tests) | days 1-15

SECONDARY OUTCOMES:
pharmacokinetics of alternative formulations | days 1-15

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1351002&StudyName=Group%20Study%20To%20Investigate%20The%20Safety%2C%20Toleration%20And%20Pharmacokinetics%20Of%20Multiple%20Oral%20Doses%20Of%20PF-04531083%20In%20Healthy%20Subjects